CLINICAL TRIAL: NCT00499070
Title: TCR Vbeta Repertoire and PNH Clones in Children With Refractory Cytopenia (RC). An Open Nonrandomised Multi-Center Prospective Study
Brief Title: Assessing Immune Function in Young Patients With Cytopenia That Did Not Respond to Treatment
Status: Completed | Type: Observational
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Charlotte Niemeyer, MD, MD Prof. Dr. med. Niemeyer, University Hospital Freiburg
Other Study IDs: CDR0000553058; EWOG-MDS-RC-06 (Other: University Hospital Freiburg)
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Dyskeratosis Congenita; Fanconi Anemia; Myelodysplastic Syndromes; Pearson Marrow-pancreas Syndrome; Shwachman-diamond Syndrome
Keywords: refractory cytopenia with multilineage dysplasia; aplastic anemia; Fanconi anemia; dyskeratosis congenita; Shwachman-Diamond syndrome; Pearson marrow-pancreas syndrome
MeSH Terms: conditions — Dyskeratosis Congenita; Fanconi Anemia; Myelodysplastic Syndromes; VLCAD deficiency; Shwachman-Diamond Syndrome; Anemia, Aplastic | interventions — Polymerase Chain Reaction; Flow Cytometry; Immunologic Techniques; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone Marrow Peripheral blood cells
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: polymerase chain reaction
Other: flow cytometry — For analyzing GPI deficient clones full blood will be analyzed by phenotyping using flowcytometry. For that purpose CD14, CD16 and CD24 expression will be evaluated in CD45 positive cells. Erythroid cells will be evaluated for CD55 and CD59 expression searching for clear populations with a lack of GPI-linked molecules. In addition, immunophenotyping using flowcytometry will be performed to evaluate which differentiation stages of the major hematopoietic lineages in BM and PB are associated with TCRVβ repertoire skewing. Comparison between BM and PB will identify which is the optimal compartment to analyze the responsible hematopoietic clones.
Other: immunologic technique
Procedure: biopsy

SUMMARY:
RATIONALE: Studying biopsy, bone marrow, and blood samples from patients with cytopenia that did not respond to treatment may help doctors learn more about the disease and plan the best treatment.

PURPOSE: This laboratory study is assessing immune function in young patients with cytopenia that did not respond to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the value of TCR V beta repertoire analysis for the determination of autoimmunity in refractory cytopenia (RC).
* To evaluate which immunophenotypic hematopoietic subclones are associated with oligoclonal T-cell expansion in RC.
* To evaluate the presence of paroxysmal nocturnal hemoglobinuria (PNH) clones in RC.

Secondary

* To compare the molecular response with the hematologic response in patients with RC after treatment with immunosuppressive therapy (IST).
* To compare the molecular response with human leukocyte histocompatability antigen (HLA) expression in patients with RC after treatment with IST.

OUTLINE: This is an open-label, multicenter, nonrandomized, prospective study.

Patients undergo biopsy, bone marrow, and blood sample collection periodically for immunological studies. Samples are analyzed for TCR V beta repertoire and paroxysmal nocturnal hemoglobinuria (PNH) clone analysis via PCR heteroduplex analysis and immunophenotyping of CD14, CD16 , CD55, CD59, and CD24 expression via flow cytometry.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of refractory cytopenia (RC) including any of the following:

  * Severe aplastic anemia (SAA)
  * Fanconi's anemia
  * Shwachman Diamond syndrome
  * Dyskeratosis congenita
  * Pearson syndrome
* All RC patients included in the EWOG MDS 2006 protocol irrespective of therapy
* Patients who have undergone hematopoietic stem cell transplantation (HSCT) may be enrolled on EWOG-MDS SCT RC RIC 06 or EWOG-MDS SCT MDS 06 protocol

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* No prior immunosuppressive therapy for refractory cytopenia

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients with MDS
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2007-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with TCR V beta oligoclonality at diagnosis | 96 months
Immunophenotype of patients with oligoclonal T-cell expansion | 96 months
Number of patients with glycophosphatidylinositol (GPI) deficient clones | 96 months

SECONDARY OUTCOMES:
Number of patients with molecular response as compared to hematological response after IST | 96 months
Number of patients with HLA-DR15 antigen expression and molecular response as compared to number of patients with other HLA-DR antigens and molecular response | 96 months
Overall survival | 96 months
Failure-free survival | 96 months

CONTACTS AND LOCATIONS:
Overall Officials: Marry M. Van Den Heuvel-Eibrink, MD, PhD, Study Chair — Erasmus MC-Sophia Children's Hospital
Locations (10):
- St. Anna Children's Hospital, Vienna, Austria
- Ghent University, Ghent, Belgium
- University Hospital Motol, Prague, Czechia
- Arhus Universitetshospital - Skejby, Aarhus, Denmark
- Universitaetskinderklinik - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Germany
- Our Lady´s Hospital for Sick Children, Dublin, Ireland
- Fondazione I.R.C.C.S. Policlinico San Matteo, Pavia, Italy
- Erasmus MC - Sophia Children's Hospital, Rotterdam, Netherlands
- Hospital Sant Joan de Deu, Barcelona, Spain
- University Children's Hospital, Zurich, Switzerland

REFERENCES:
- [Derived] Aalbers AM, van den Heuvel-Eibrink MM, Baumann I, Dworzak M, Hasle H, Locatelli F, De Moerloose B, Schmugge M, Mejstrikova E, Novakova M, Zecca M, Zwaan CM, Te Marvelde JG, Langerak AW, van Dongen JJ, Pieters R, Niemeyer CM, van der Velden VH. Bone marrow immunophenotyping by flow cytometry in refractory cytopenia of childhood. Haematologica. 2015 Mar;100(3):315-23. doi: 10.3324/haematol.2014.107706. Epub 2014 Nov 25. PMID 25425683
- [Derived] Aalbers AM, van den Heuvel-Eibrink MM, Baumann I, Beverloo HB, Driessen GJ, Dworzak M, Fischer A, Gohring G, Hasle H, Locatelli F, De Moerloose B, Noellke P, Schmugge M, Stary J, Yoshimi A, Zecca M, Zwaan CM, van Dongen JJ, Pieters R, Niemeyer CM, van der Velden VH, Langerak AW. T-cell receptor Vbeta skewing frequently occurs in refractory cytopenia of childhood and is associated with an expansion of effector cytotoxic T cells: a prospective study by EWOG-MDS. Blood Cancer J. 2014 May 2;4(5):e209. doi: 10.1038/bcj.2014.28. PMID 24786393